CLINICAL TRIAL: NCT05420818
Title: Does Inversion and Fixation of the Transversalis Fascia Prevent Postoperative Seroma Formation in Patients Undergoing Laparoscopic Inguinal Hernia Repair?
Brief Title: Inversion and Fixation of the Transversalis Fascia in Laparoscopic Inguinal Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erol Aydın, MD, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2983
Record Dates: First submitted 2022-05-13; First posted 2022-06-15 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Hernia, Inguinal
Keywords: Inguinal Hernia; TEP; Seroma; Laparoscopic Hernia; Transversalis fascia inversion
MeSH Terms: conditions — Hernia, Inguinal; Seroma | interventions — tetraethylpyrazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Experimental): Patients who underwent transversalis fascia inversion during TEP
  Interventions: Procedure: Transversalis Fascia Inversion
- Control Group (No Intervention): Patients who did not undergo transversalis fascia inversion during TEP

INTERVENTIONS:
Procedure: Transversalis Fascia Inversion — This study will be carried out at SBU Istanbul Training and Research Hospital, General Surgery Clinic. Patients diagnosed with M2 and M3 direct primary inguinal hernia according to EHS classification and who will undergo TEP repair surgery will be randomized into 2 groups. After direct hernia reduction in the patients in the first group, the transversalis fascia at the hernia site will be pulled inward and fixed to the Cooper ligament with 2 or 3 absorbable tackers. Standard surgery will then be continued. The patients in the second group will undergo standard surgery without any seroma prevention procedure. Demographic data of patients in both groups, postoperative pain (VAS values) at postoperative 1st, 7th day and 3rd month, clinical/radiological seroma rate, postoperative pain, QOL, recurrence and other complications will be recorded. When the desired number of patients and follow-up period are reached, the data in the 2 groups will be compared.
  Other Names: TEP
  Arms: Active Group

SUMMARY:
According to the EHS classification, at least 80 patients who will undergo TEP repair for the first time with the diagnosis of M2 and M3 direct inguinal hernia will be randomized into 2 groups. After direct hernia reduction in the patients in the first group, the transversalis fascia at the hernia site will be pulled inward and fixed to the Cooper ligament with 2 or 3 absorbable tackers. Standard surgery will then be continued. The patients in the second group will undergo standard surgery without any seroma prevention procedure. Demographic data, clinical/radiological seroma rate, postoperative pain (VAS values),quality of life(SF36 questionnaire), recurrence and other complications at postoperative 1st, 7th day, 3rd and 6th month will be monitored. When the desired number of patients and the follow-up period are reached, the data in the 2 groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or/and radiological diagnosis of primary inguinal hernia
* EHS type M2 and M3 direct hernias
* Laparoscopic totally extraperitoneal (TEP) repair

Exclusion Criteria:

* Indirect hernias
* M1 direct hernias
* Recurrent hernias
* Patients with previous groin operations on same side
* Pregnant women
* Patients who did not accept to participate in the study
* ASA score of 3 or higher,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-05-05 (Estimated); Study Completion 2023-07-05 (Estimated)

PRIMARY OUTCOMES:
Seroma formation rate | 3 month
  The clinical/radiological seroma formation rates between the groups with and without transversalis fascia inversion and fixation.

SECONDARY OUTCOMES:
Chronic pain and quality of life measures | 3 month
  Detect the presence of chronic pain and measuring quality of life after 3 months using the SF-36
Pain levels | 7 day
  Pain Scores on the Visual Analog Scale at postoperative 7tht day
Postoperative pain levels | 1 day
  Pain Scores on the Visual Analog Scale at postoperative 1st day

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Research and Training Hospital, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided